CLINICAL TRIAL: NCT03716336
Title: Impact of Concurrent Aerobic and Strength Training With Caloric Restriction on Insulin Resistance in Obese Premenopausal Women: A Randomized Controlled Trial
Brief Title: Aerobic and Strength Training With Caloric Restriction on Insulin Resistance in Obese Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor of physical therapy for women's health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU90
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Insulin Resistance Syndrome
Keywords: resistive exercises; aerobic exercises; diet; insulin resistance; premenopausal
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Resistance Training; Exercise

STUDY DESIGN:
Intervention Model Description: were randomly assigned to group A participated in aerobic and resistive exercise program, and group B participated in aerobic exercise and followed prescribed diet restriction program. Both of the groups (A&B) followed the treatment program 3 times per weeks for 8 weeks. Assessment of the fasting glucose, fasting insulin, and HOMA test of insulin resistance were measured for all subjects in both groups (A and B) was carried out before and after the end of the treatment program.
Who Masked: Outcomes Assessor
Masking Description: Participants were assigned randomly used sealed envelope into two groups (A&B) equally in number.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise (Other): walking on treadmill
  Interventions: Other: Resistance exercise; Other: Aerobic exercise; Dietary Supplement: diet restriction
- resistive exercise (Other): Resistance exercise were performed for all participants in group (A) included 9 exercise for big muscles of upper limbs
  Interventions: Other: Resistance exercise; Other: Aerobic exercise; Dietary Supplement: diet restriction

INTERVENTIONS:
Other: Resistance exercise — Resistance exercise were performed for all participants in group (A) only included 9 exercise for big muscles of upper limbs (shoulder flexors muscles, shoulder extensors and shoulder abductors), lower limbs (hip flexors, hip extensors and knee flexors and knee extensors) and abdominal muscle using moderate work load (60 - 75% of IRM) 1set of 10 repetitions, progressing to 2 sets of 10 repetitions after four weeks for 20 minutes
Other: Aerobic exercise — aerobic exercise were performed on treadmill. For 20 minutes. All patients in both groups (A,B) had attended the program of a resistance exercises and followed by aerobic exercise for 8 weeks in form of 20 minutes walking on the treadmill without inclination.
  Other Names: exercise
Dietary Supplement: diet restriction — All participants in both groups (A,B) were instructed to follow a moderate restricted diet limited to (1800-2000) kcal/ day under supervision of a certified dietician. The diet contained: Protein and fibers: 20% carbohydrate: 50-60%, fat: low 20%.

SUMMARY:
A total of 42 premenopausal women diagnosed clinically as having insulin resistance. Their ages ranged from 35 to 45 years old; their body mass index was >30 kg/m2 and They were obese women complained of insulin resistance and non diabetic or cardiovascular disease, were randomly assigned to group A participated in aerobic & resistive exercise program, and group B participated in aerobic exercise and followed prescribed diet restriction program. Both of the groups (A&B) followed the treatment program 3 times per weeks for 8 weeks. Assessment of the fasting glucose, fasting insulin, and HOMA test of insulin resistance were measured for all subjects in both groups (A and B) was carried out before and after the end of the treatment program

DETAILED DESCRIPTION:
Forty two obese premenopausal women diagnosed as having insulin resistance were participated in this study. They were selected randomly from the out Patient Clinic of Obstetrics at Kasr El Ainy University Hospital, Faculty of Medicine, Cairo University. Their age ranged from 35 - 45years, their body mass (BMI) were>30kg/m2. Exclusion criteria of the study were as follows: Patients having diabetic or cardiovascular disease, Patients with life threatening disorders as renal failure and myocardial infarction, Patients with active malignancy and patients with severe hemorrhage, hyperthyroidism, acute viral diseases and mental disorders. Participants were assigned randomly used sealed envelope into two groups (A&B) equally in number. Group (A): (Combined resistive and aerobic exercise group) consisted of 20 women were participated in aerobic & resistive exercise program plus diet restriction, 3 times per weeks for 8 weeks. Group (B): consisted of 20 women were participated in aerobic exercise plus diet restriction 3 times per weeks for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Their age ranged from 35 - 45years.
* their body mass (BMI) were>30kg/m2.

Exclusion Criteria:

* Patients having diabetic or cardiovascular disease.
* Patients with life threatening disorders as renal failure and myocardial infarction
* Patients with active malignancy.
* patients with severe hemorrhage
* hyperthyroidism.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
HOMA test of insulin | 8 weeks
  A sample of 5ml of venous blood sample was drawn from the ante cubital vein after 10 hours fasting from all women in the two groups (A, B) for measurement of fasting blood glucose, fasting blood insulin and detection of insulin resistance (by HOMA-IR)

SECONDARY OUTCOMES:
fasting blood insulin level | 8 weeks
  A sample of 5ml of venous blood sample was drawn from the ante cubital vein after 10 hours fasting from all women in the two groups (A, B) for measurement of fasting blood insulin
fasting blood glucose level | 8 weeks
  A sample of 5ml of venous blood sample was drawn from the ante cubital vein after 10 hours fasting from all women in the two groups (A, B) for measurement of fasting blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — institutional review board of the Faculty of physical therapy, Cairo University
Locations (1):
- Faculty of physical therapy- Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No